CLINICAL TRIAL: NCT03560375
Title: The Effect of a Circuit Resistance Training, Empagliflozin or "Vegeterranean Diet" on Physical and Metabolic Function in Elderly Subjects With Type 2 Diabetes: a Study Protocol for a Randomized Control Trial (CEV-65 Trial)
Brief Title: Mediterranean Diet, Circuit Resistance Training, Empagliflozin in Elderly With Type 2 Diabetes: a Study Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLV-0816-17
Record Dates: First submitted 2018-05-06; First posted 2018-06-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2; Sarcopenia; Weight Loss
Keywords: Type 2 diabetes; Sarcopenia; Weight loss; Physical function; Metabolic control; Older adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia; Weight Loss | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label (primary outcome assessors blinded), parallel group, clinical trial of circuit resistance training for 10 weeks; V-Med diet for 10 weeks and then circuit resistance training on top of diet for 10 weeks; empagliflozin 10mg/day for 10 weeks and then circuit resistance training on top of drug therapy for 10 weeks in subjects with type 2 diabetes mellitus
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment and blinding of primary outcome assessors will be implemented
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Circuit resistance training (CRT) (Experimental): 2-3 circuits * 10 exercises * 3 times per week
  Interventions: Behavioral: Circuit resistance training (CRT)
- Empagliflozin 10 MG (Experimental): 10 mg once daily
  Interventions: Drug: Empagliflozin 10 MG
- Vegeterranean diet (V-Med diet) (Experimental): The modified V-Med diet will be considered as ad-libitum (using fat sources), aimed for sufficient protein from animal and mainly plant-based sources with carbohydrates limitation.
  Interventions: Behavioral: Vegeterranean diet (V-Med diet)

INTERVENTIONS:
Behavioral: Circuit resistance training (CRT) — Subjects will be allocated to CRT which consists of 10 resistance exercises for different body parts (=1 circuit) repeated 12-15 times, using modest weights (approximately 40-60% of one repetition maximum, RM). Each exercise is expected to be completed within 30-40 sec. The participant will move quickly (within 15-30 seconds) from one exercise to the next. The circuit will be repeated up to three times depending on the week of intervention. Thus, it will take about 30 min to complete an exercise session. For a summary of articles on CRT in older adults based on a meta-analysis, we performed please see:
  Circuit resistance training is an effective means to enhance muscle strength in older and middle-aged adults: A systematic review and meta-analysis. Ageing Res Rev. 2017 Aug;37:16-27
  Arms: Circuit resistance training (CRT)
Behavioral: Vegeterranean diet (V-Med diet) — The modified V-Med diet will be considered as ad-libitum (using fat sources) aimed for a minimum of 1 gr/kg/day of protein, limiting carbohydrates: 3 servings for men and 2 servings for women per main meal and 1 serving per intermediate meal for both genders. Subjects will be asked to avoid red meat and poultry completely and the consumption of dairy and eggs products will be limited to 2 servings per day. 2-3 servings of fish should be consumed during the week. The rest of protein consumption will be recommended from legumes sources. The target legume consumption will be 1.5 cup per day (2 servings per day) of cooked beans, chickpeas, lentils and/or using pulses-based flour or pulses-based bread. Consumption of whole grain carbohydrate foods will be recommended.
  Arms: Vegeterranean diet (V-Med diet)
Drug: Empagliflozin 10 MG — Subjects allocated to empagliflozin will be asked to add empagliflozin 10mg, preferably in the morning, to their medication regimen. Subjects will be monitored for adverse events including hypoglycemic events during all study visits.
  Arms: Empagliflozin 10 MG

SUMMARY:
Primary objective: To assess the effects of a modified plant-based Mediterranean diet (vegeterranean diet), circuit resistance training (CRT) and empagliflozin alone or in combination on metabolic and physical function in elderly subjects with type 2 diabetes. The rationale for this study is to assess three interventions associated with a negative energy/caloric balance (increased caloric use in exercise, caloric restriction in the vegeterranean diet and caloric wasting by glycosuria with empagliflozin), their interaction and effect on body composition and physical function.

Methods and analysis: One hundred men and women ≥ 65 years of age with type 2 diabetes, and low levels of physical activity will be randomized (1:1:1 manner, gender-stratified) for 10 weeks to one of 3 parallel arms: CRT consisting of 3 home sessions/week; ad-libitum plant-based Mediterranean diet (limited consumption of eggs, dairy and fish, avoidance of red meat and poultry) or empagliflozin 10mg/day. After 10 weeks CRT will be added to the empagliflozin or diet arms for an additional 10 weeks. Allocation concealment and blinding of primary outcome assessors will be implemented. Efficacy will be determined by assessment of lean body mass, body weight, fat mass %, sarcopenia measures (such as strength and physical function), HbA1c and blood pressure as well as other outcomes (both objective and subjective). Safety will be evaluated by routine monitoring of adverse events. This study was approved by the Tel-Aviv Sourasky Medical Center Institutional Review Board

ELIGIBILITY:
Inclusion Criteria:

Subjects who have type 2 diabetes mellitus in accordance with American Diabetes Association guidelines and:

1. Are ≥65 years of age (inclusive) on the day of signing the informed consent form.
2. Perform <2 days a week of any leisure aerobic physical activity (PA), who are able to walk independently either with or without an assistance device (cane or walker).
3. HbA1C ≥6.5% to ≤8%.

Exclusion Criteria:

1. Recent use of steroid agents (<6 months, replacement therapy is allowed)
2. Uncorrected hypothyroidism [thyroid stimulating hormone (TSH) > 6 mlU/L]
3. Diagnosis of malignancy within the past 5 years except for non-melanoma skin cancer.
4. Severe kidney disease (eGFR<45cc/ml)
5. Active depression
6. Recent (≤6 months) or unstable cardiovascular condition; New York Heart Association (NYHA) Class 3 or higher congestive heart failure;
7. Subjects with PA limiting pain due to neuropathy
8. Subjects who are in an active nutritional therapy changed their diet recently (<1 month) and/or in a weight-loss program (actively losing weight).
9. Has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
A composite of metabolic and functional indices | After 10 weeks (for all 3 arms) and after 20 weeks (for diet and drug arms only)
  In the 'metabolic index' 1 point was given for achieving a reduction of at least 2% in body fat, 2cm of waist circumference, 0.5% HbA1c and 5mmHg systolic blood pressure (final score 0-4). Metabolic threshold values that reflect the desired reduction were chosen based preferably on meta-analyses of randomized trials (or single RCT) that examined the impact of weight loss/lifestyle interventions (diet and/or physical exercise - focus on interventions as similar to our interventions) and pharmacotherapy (e.g., empagliflozin) in populations of overweight and obese (with/without diabetes) adults/ older adults. We reviewed the threshold values and set the final values taking into account the data reviewed for each metabolic variable.The 'functional index' awarded one point for preservation or increase in total skeletal muscle mass, HGS, isometric knee extension, and TUG results (final score 0-4).

SECONDARY OUTCOMES:
Change in fasting plasma glucose | After 10 weeks (for all 3 arms) and after 20 weeks (for diet and drug arms only)
  Change in fasting plasma glucose (%) will be calculated as fasting plasma glucose (mg/dl) at the end of 10 weeks (and 20 weeks) minus baseline fasting plasma glucose divided by fasting plasma glucose at baseline and multiplied by 100.
Change in sarcopenia | After 10 weeks (for all 3 arms) and after 20 weeks (for diet and drug arms only)
  Sarcopenia will be assessed by results obtained in the In-Body (720) body composition analyzer, following the consensus definitions offered elsewhere (Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, et al. Sarcopenia: European consensus on definition and diagnosis. Age Ageing. 2010 Jul;39(4):412-23.). Shortly, the skeletal muscle index (SMI = skeletal muscle mass/body mass x 100) will be compared to gender-specific reference norms of young adults (aged 18-39 years). Sarcopenia will be defined as any value < 10.76 kg/m2 for men and < 6.76 kg/m2 for women. Sarcopenia change will be considered as "improved vs. not improved"; change from one level to the other
Change in strength | After 10 weeks (for all 3 arms) and after 20 weeks (for diet and drug arms only)
  Grip strength, assessed as the average of 3 readings of the dominant hand by a handheld dynamometer [Jamar® Plus+ Digital Hand Dynamometer (Jamar® Smart) 200-lb.]. Change in grip strength (%) will be calculated as grip strength at the end of 10 weeks (and 20 weeks) minus baseline grip strength divided by grip strength at baseline and multiplied by 100.
Relative lean mass change | after 10 weeks (for all 3 arms) and after 20 weeks (for diet and drug arms only)
  Relative lean mass change will be calculated as % lean mass (the proportion of lean mass out of weight) at the end of study minus % lean mass at baseline divided by lean mass % at baseline and multiplied by 100

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute of Endocrinology Metabolism and Hypertension, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kis O, Buch A, Eldor R, Rubin A, Dunsky A, Stern N, Moran DS. Should knee extension strength testing be implemented as a screening test for identifying probable and confirmed sarcopenia in older T2DM patients? Eur Rev Aging Phys Act. 2022 Jan 27;19(1):5. doi: 10.1186/s11556-021-00280-y. PMID 35086483
- [Derived] Buch A, Eldor R, Kis O, Keinan-Boker L, Dunsky A, Rubin A, Lopez A, Sofer Y, Osher E, Marcus Y, Stern N. The effect of circuit resistance training, empagliflozin or "vegeterranean diet" on physical and metabolic function in older subjects with type 2 diabetes: a study protocol for a randomized control trial (CEV-65 trial). BMC Geriatr. 2019 Aug 22;19(1):228. doi: 10.1186/s12877-019-1219-7. PMID 31438863